CLINICAL TRIAL: NCT05561816
Title: Opened, Multicenter, Randomized, in Parallel Groups Comparative Study to Assess Efficacy and Safety of Dioxidin®, Solution for Topical and External Application 0.025% (Valenta Farm, Russia) and Miramistin®, Solution for Topical Application 0.01% (Infamed K LLC, Russia) in Treatment of Superficial Pyoderma
Brief Title: Efficacy and Safety of Dioxidin Versus Miramistin in Superficial Pyoderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIO-09-2020
Record Dates: First submitted 2022-09-15; First posted 2022-09-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pyoderma
MeSH Terms: conditions — Pyoderma | interventions — miramistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dioxidin (Experimental): Patients will apply Dioxidin® 3 times a day (in the morning, afternoon and evening) by spraying (4 pressings of the spray nozzle on each affected area corresponding to 1% of the body area) on the affected skin areas from a distance of about 10 cm, so that the entire affected surface is covered with the solution. After application, you should wait until the preparation is completely dry. The therapy duration will be 10 days.
  Interventions: Drug: Hydroxymethylquinoxalindioxyde
- Miramistin (Active Comparator): Patients will apply Miramistin® to the affected areas of the skin by wiping with sterile gauze swabs liberally moistened with the preparation three times a day (in the morning, lunchtime, and evening). The therapy duration will be 10 days.
  Interventions: Drug: Benzyl-dimethyl-[3-(tetradecanoylamino)propyl]azanium

INTERVENTIONS:
Drug: Hydroxymethylquinoxalindioxyde — Dioxidin®, 0.025% solution for local and external use (Valenta Farm, Russia).
  Other Names: Dioxidin
  Arms: Dioxidin
Drug: Benzyl-dimethyl-[3-(tetradecanoylamino)propyl]azanium — Miramistin®, topical solution 0.01% (Infamed K LLC, Russia)
  Other Names: Miramistin
  Arms: Miramistin

SUMMARY:
The study is aimed to:

* evaluate the effectiveness of 10-day therapy with Dioxidin® compared with Miramistin® in the treatment of superficial pyoderma,
* evaluate the safety and tolerability of 10-day therapy with Dioxidin® compared with Miramistin® for the treatment of superficial pyoderma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 years inclusive.
2. Signed informed consent form to participate in the study.
3. Patients with superficial pyoderma of different localization.
4. Body surface lesion area ≤ 5%.
5. Patient's willingness and ability to comply with protocol requirements throughout the study (in particular, willingness to adhere strictly to the prescribed treatment regimen and to record the time of drug administration in the patient's diary).
6. Consent of study participant with preserved reproductive potential to use adequate methods of contraception (e.g., dual barrier method) throughout the study and for 3 weeks after study completion.

Exclusion Criteria:

1. Hypersensitivity to the active and/or excipients of the studied drugs.
2. Presence of signs of acute respiratory infections.
3. Deep pyoderma (furunculus, carbuncle, abscess, hydradenitis, etc.).
4. Use of local and systemic antibacterials, antiseptics, glucocorticosteroids, and antifungal agents less than 14 days prior to the screening visit.
5. Presence of infectious diseases requiring topical and/or systemic antibacterial therapy.
6. Vaccination of the patient less than 1 week prior to the screening visit.
7. Adrenal insufficiency.
8. Body temperature >37C.
9. Fungal, viral skin infections, severe generalized bacterial skin lesions, other skin diseases.
10. Immunodeficiency states.
11. Positive HIV, Hepatitis B and C, or syphilis, or SARS-CoV-2 rapid test (COVID-19)
12. Presence of at least one of the following epidemiologic indicators: Return from foreign travel 7 days prior to screening; Close contact in the last 7 days prior to screening with an individual under observation for COVID-19 who subsequently became ill; Close contact in the last 7 days prior to screening with an individual with a laboratory confirmed diagnosis of COVID-19; Professional contacts in the last 7 days prior to screening with individuals who have a suspected or confirmed case of COVID-19.
13. Scalp lesion (where treatment procedures and effectiveness cannot be adequately evaluated due to thick/long hair).
14. Allergic reactions to antibacterial drugs, antiseptic drugs in history.
15. Diabetes mellitus type 1 or 2.
16. Any other comorbidities or conditions that, in the opinion of the investigator, make it difficult to interpret treatment results or make it impossible to perform procedures in this clinical trial or pose a risk to the patient when participating in the study (e.g., a history of severe allergies, atopic dermatitis in case the affected area overlaps with the area of pyoderma).
17. History of malignancy, with the exception of patients who have not had the disease in the past 5 years, patients with fully cured basal cell carcinoma of the skin, or fully cured carcinoma in situ.
18. Severe, decompensated, or unstable somatic diseases (any disease or condition that is life-threatening or worsens the patient's prognosis, or makes it impossible for the patient to participate in a clinical trial).
19. The need for concomitant therapy with any of the drugs listed as "Prohibited Concomitant Treatment".
20. History of alcohol and/or drug dependence.
21. Participation in another clinical trial less than 3 months prior to the Screening Visit.
22. Pregnancy.
23. Breastfeeding period.

Withdrawal Criteria:

1. Withdrawal of Informed Consent by the patient.
2. Patient does not meet inclusion criteria.
3. Patient is found to have non-inclusion criteria.
4. Patient's desire to stop their participation in the study at any stage of the study.
5. Researcher's decision that continued participation in the study is contrary to the patient's best interests.
6. The investigator's decision to exclude the patient from the study due to a serious deviation from/breach of protocol.
7. Identification of a probable or confirmed COVID- 19 case (according to the Standard COVID-19 case definition).
8. An undesirable event requiring withdrawal of study therapy, or prescription of drugs from the Prohibited Complementary Treatment section, or limiting protocol procedures.
9. Patient's failure to show up for any visit and loss of communication with the patient.
10. Patient's omission of a cumulative total of more than 5 doses of medication throughout the treatment period or 3 consecutive doses.
11. Pregnancy.
12. Termination of the study by the sponsor.
13. Termination of the study by the investigator.
14. Termination of the study by the regulatory agency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experienced complete cure of the disease at Visit 4 | Day 10
  In this study, cure will be considered achieved if the severity of each pyoderma symptom (painfulness on palpation, pustules/fluketens, hyperemia, inflammatory infiltration, edema) does not exceed 0 points (assessed from 0 [the absence of symptom] to 3 [maximal severity of the symptom])

SECONDARY OUTCOMES:
Mean change in the arithmetic mean change in pyoderma symptom severity scale, to Visits 2, 3, and 4 compared to baseline. | Day 1, Day 4, Day 7, Day 10
  Each symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Mean change in severity for the symptom "soreness on palpation" to Visits 2, 3 and 4 compared to baseline | Day 1, Day 4, Day 7, Day 10
  The symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Average change in the severity for the symptom "presence of pustules/flukteness" to Visits 2, 3 and 4 compared to baseline | Day 1, Day 4, Day 7, Day 10
  The symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Average change in the expression for the symptom "hyperemia" to Visits 2, 3 and 4 compared to baseline | Day 1, Day 4, Day 7, Day 10
  The symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Mean change in severity for the symptom "inflammatory infiltration" to Visits 2, 3 and 4 compared to baseline | Day 1, Day 4, Day 7, Day 10
  The symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Mean change in severity for the symptom "swelling" to Visits 2, 3 and 4 compared to baseline | Day 1, Day 4, Day 7, Day 10
  The symptom will be assessed from 0 (the absence of symptom) to 3 (maximal severity of the symptom)
Average patient satisfaction with treatment at Visit 2, 3 and 4 | Day 4, Day 7, Day 10
  The satisfaction will be assessed from 0 (not satisfied) to 3 (absolutely satisfied)
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, Day 1, Day 4, Day 7, Day 10
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, Day 1, Day 4, Day 7, Day 10
  DBP, mmHg
Safety and Tolerability: vital signs - heart rate (HR) | Screening, Day 1, Day 4, Day 7, Day 10
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, Day 1, Day 4, Day 7, Day 10
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, Day 1, Day 4, Day 7, Day 10
  Physical examination will follow the general rules of internal medicine: general examination, examination of mucous membranes and skin, including palpation of lymph nodes, evaluation of the musculoskeletal system, palpation, percussion, and auscultation of the main organ systems (cardiovascular, respiratory, digestive, and urinary systems) will be performed sequentially. The findings (if any) will be reported as the rate of clinically significant findings by each system level assessed.
Safety and Tolerability: complete blood count - hemoglobin | Screening, Day 10
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, Day 10
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, Day 10
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, Day 10
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, Day 10
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, Day 10
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - lymphocytes | Screening, Day 10
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, Day 10
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, Day 10
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, Day 10
  Basophils, %
Safety and Tolerability: complete blood count - neutrophils | Screening, Day 10
  Neutrophils, % (segmented and stab)
Safety and Tolerability: blood test results - glucose | Screening, Day 10
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, Day 10
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening, Day 10
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total protein | Screening, Day 10
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening, Day 10
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - urea | Screening, Day 10
  Urea in blood serum, mmol/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, Day 10
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, Day 10
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, Day 10
  ALP in blood serum, U/L
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 10
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, Day 10
  Color of the urine, visual assessment (pale yellow, yellow, amder, brown etc.)
Safety and Tolerability: urinalysis - transparency | Screening, Day 10
  Transparency of the urine, visual assessment (transparent or cloudy)
Safety and Tolerability: urinalysis - pH | Screening, Day 10
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, Day 10
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 10
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, Day 10
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, Day 10
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - epithelial cells | Screening, Day 10
  Epithelial cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders | Screening, Day 10
  Cylinders in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, Day 10
  Bacteria in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - mucus | Screening, Day 10
  Presence of mucus in the urine
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study (Day 17)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: local reactions | From the date of screening (and signing informed consent form) to the end of the study (Day 17)
  Local reactions at the site of application will be evaluated separately on a 4-point scale (0 - no local reaction, 1 - weak local reaction in a limited area at the site of application, 2 - moderate local reaction in a limited/all area of application, 3 - strong local reaction in the whole area of application or going beyond it)

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Chelyabinsk Regional Clinical Dermatology and Venereology Dispensary, Chelyabinsk
  - Professor Gorbakov Clinic, LLC, Krasnogorsk
  - Moscow Scientific and Practical Center of Dermatovenerology and Cosmetology of the Moscow Department of Health, Moscow
  - Federal State Budgetary Educational Institution of Higher Professional Education Ryazan State Medical University, Ministry of Health of Russia, Ryazan
  - Regional Clinical Dermatology and Venereology Dispensary, Ryazan
  - City Dermatological and Venereological Dispensary, Saint Petersburg
  - Northwestern Center for Evidence-based Medicine, JSC, Saint Petersburg
  - Private Health Care Institution "Clinical Hospital "RZD-Medicine" of St. Petersburg, Saint Petersburg
  - Yakusi Clinic, LLC, Saint Petersburg
  - Clinic of Modern Medicine of Dr. Bogorodskaya, LLC, Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided